CLINICAL TRIAL: NCT04970043
Title: A Single Arm, Prospective, and Exploratory Clinical Study of Camrelizumab Combined With Pemetrexed and Carboplatin in Advanced Non-small Cell Lung Cancer Patients With EGFR Mutation Who Failed EGFR-TKI Treatment
Brief Title: Camrelizumab Combined With Pemetrexed and Carboplatin for the Study of EGFR-mutated Lung Squamous NSCLC Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN, Assistant Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJ-NSCLC-IIT-Camrelizumab
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Lung Cancer Stage II
Keywords: Non-small Cell Lung Cancer; PD-1 Antibody
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+ pemetrexed + platinum (Experimental)
  Interventions: Drug: Camrelizumab+ pemetrexed + platinum

INTERVENTIONS:
Drug: Camrelizumab+ pemetrexed + platinum — Induction period: (4-6 cycles) Camrelizumab: a fixed dose of 200 mg, intravenous drip for 30-60 minutes, the first day, every 3 weeks as a cycle.
  Pemetrexed: 500 mg / m2, given on the first day, every 3 weeks as a cycle; Carboplatin: AUC = 4-5, given on the first day, every 3 weeks as a cycle; After 4-6 cycles of treatment, the patients entered the maintenance treatment period of carrizumab combined with pemetrexed.
  Maintenance treatment period:
  Camrelizumab: a fixed dose of 200 mg, intravenous drip for 30-60 minutes, the first day, every 3 weeks as a cycle.
  Pemetrexed: 500 mg / m2, given on the first day, every 3 weeks as a cycle; Every 3 weeks is a treatment cycle, and the drug is maintained until the following conditions occur: disease progression, intolerable toxicity, or receiving immunotherapy for no more than 35 cycles (2 years).

SUMMARY:
A single-arm, prospective, single-center, phase II, exploratory study investigating Camrelizumab combined with pemetrexed and carboplatin in the treatment of advanced non-squamous cell non-small-scale EGFR mutations (EGFR-TKI treatment failure ) Effectiveness of cell lung cancer patients

DETAILED DESCRIPTION:
In this study, eligible subject will be Subjects will have the opportunity to receive the treatment of Camrelizumab in combination with pemetrexed and carboplatin therapy .

ELIGIBILITY:
Inclusion Criteria:

* 1. The age is 18-70 years old;

  2. According to the TNM staging of lung cancer in the 8th edition of the International Association for the study of lung cancer and the Joint Committee on American Classification of cancer, non squamous non-small cell lung cancer confirmed by histology or cytology that can not be treated surgically and can not receive radical concurrent chemoradiotherapy and locally advanced or metastatic (stage Ⅲ B, Ⅲ C or Ⅳ) non squamous non-small cell lung cancer;

  3. EGFR mutation (deletion of exon 19 and L858R mutation of exon 21) was confirmed by tumor histology, cytology or hematology before EGFR / - TKI treatment;

  4. After EGFR-TKI treatment failure (based on RECIST v1.1, disease progression confirmed by imaging), it meets any of the following requirements:
  1. In the past, the first or second generation EGFR-TKI (such as icotinib, gefitinib, erlotinib, afatinib or other first or second generation EGFR-TKI listed in China) failed, and the T790M mutation of EGFR 20 exon should be confirmed by histology;
  2. In the past, he received the first or second generation EGFR-TKI (e.g. icotinib, gefitinib, erlotinib, afatinib), and the T790M mutation of EGFR 20 exon was confirmed by histology or hematology during or after the treatment failure. Then he received the third generation EGFR-TKI (e.g. oxitinib or other third-generation EGFR-TKI listed in China) and failed;
  3. The patients who received the third-generation EGFR-TKI (such as oxitinib or other third-generation EGFR-TKI listed in China) at the time of initial diagnosis of EGFR mutant NSCLC and progressed without other targeted treatment opportunities;

  5. No previous systemic anti-tumor therapy (except EGFR-TKI) for advanced non squamous NSCLC (for those who have received platinum neoadjuvant chemotherapy or adjuvant chemotherapy, if the disease progression occurred more than 6 months after the end of the last treatment, they are eligible to participate in this study);

  6. The life expectancy is at least 3 months;

  7. ECoG score: 0-1;

  8. According to recist1.1, the researcher confirmed that there was at least one measurable lesion;

  9. The function of main organs is normal, and the test results must meet the following requirements:
  1. The standard of blood routine examination should be met (no blood transfusion and blood products within 14 days, no correction with G-CSF and other hematopoietic stimulating factors)

     A. Hemoglobin (HB) ≥ 90 g / L;

     B. Neutrophil count (ANC) ≥ 2 × 109/L；

     C. Platelet count (PLT) ≥ 100 × 109/L；
  2. Biochemical tests should meet the following standards:

     A. Total bilirubin (TBIL) < 1.5 upper limit of normal (ULN);

     B. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5uln, but < 5uln for patients with liver metastasis;

     C. Serum creatinine (CR) ≤ 1.5 ULN or endogenous creatinine clearance > 60 ml / min (Cockcroft Gault formula);

     D. Urine routine test results showed that urinary protein (Upro) < 2 + or 24-hour urinary protein < 1g;

  10. Women of childbearing age must have taken reliable contraceptive measures or conducted pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and they are willing to use appropriate contraceptive methods during the test period and 60 days after the last administration of the test drug. For men, it is necessary to agree to use appropriate contraceptive methods or surgical sterilization during the trial period and 120 days after the last administration of the trial drug;

  11. Signed the written informed consent, and expected to have good compliance with the research protocol.

Exclusion Criteria:

* 1. Patients with active brain metastases (for patients with stable symptoms of brain metastases after treatment, keep stable for at least 4 weeks);

  2. Previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that stimulate or synergistically inhibit T cell receptors (e.g., CTLA-4, OX-40, CD137);

  3. Have received systemic anti-tumor therapy (including cytotoxic chemotherapy combined with radiotherapy) for advanced NSCLC other than EGFR-TKI in the past;

  4. Immunosuppressive drugs were used within 14 days before the first use of karelizumab, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroids (i.e. not more than 10 mg / day prednisolone or other corticosteroids with the same physiological dose of drugs);

  5. Received systemic treatment of Chinese herbal medicine with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use to control pleural effusion) within 2 weeks before the first administration;

  6. Received EGFR-TKI within 2 weeks before the first administration;

  7. Received palliative radiotherapy within 7 days before the first administration. For the patients who had received palliative radiotherapy 7 days before the first administration, all the following conditions must be met before they can be enrolled: there is no toxic reaction related to radiotherapy, glucocorticoid is not required, and radiation pneumonia is excluded;

  8. Severe cardiovascular diseases: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia (including QTc interval ≥ 450 ms for male and ≥ 470 MS for female); Grade Ⅲ - Ⅳ cardiac insufficiency (according to NYHA classification of New York Heart Association, see Annex 3), or left ventricular ejection fraction (LVEF) < 50% by echocardiography;

  9. Currently participating in interventional clinical research treatment, or receiving other research drugs or research devices within 4 weeks before the first administration; Not fully recovered from toxicity and / or complications caused by any intervention before the first administration (i.e., ≤ grade 1 or baseline, excluding fatigue or hair loss);

  10. With uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (drainage once a month or more frequently);

  11. Subjects have received or plan to receive solid organ or blood system transplantation (except corneal transplantation) during the study period;

  12. Patients with active autoimmune disease or immunodeficiency, or with the above history, including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, rheumatoid arthritis, inflammatory bowel disease, hypophysitis, vasculitis, nephritis, etc.) were not included. The following exceptions: Patients with a history of autoimmune hypothyroidism but receiving thyroid hormone replacement therapy were included in the study. Patients with type 1 diabetes whose blood glucose is controlled after insulin administration can participate in this study.

  13. Subjects who received systemic therapy such as bronchodilators were not satisfied with asthma control and could not be included (those who had complete remission of asthma in childhood and did not need any intervention in adulthood could be included).

  14. Severe infection occurred within 4 weeks before the first administration (e.g. need for intravenous drip of antibiotics, antifungal or antiviral drugs), or fever of unknown origin > 38.5 ° C occurred during the screening period / before the first administration; Or received major surgical treatment within 3 weeks before the first medication;

  15. Inoculate live attenuated vaccine within 30 days of the first administration or expected during the study period;

16.16. Human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS), untreated active hepatitis B, hepatitis C virus (hepatitis C antibody positive, and HCV-RNA higher than the lower limit of analysis method) or combined hepatitis B and hepatitis C common sense;

Note: the hepatitis B subjects who met the following criteria also met the inclusion criteria: HBV viral load must be <1000 copy /ml (200 IU/ml) before the first dose, and the subjects should be treated with anti HBV therapy during the whole chemotherapy course to avoid virus reactivation. For the subjects with anti HBC (+), HBsAg (-), anti HBS (-) and HBV viral load (-), preventive anti HBV treatment is not necessary, but close monitoring of virus reactivation is needed;

17. Patients with a clear history of allergy are known to have allergic reactions to carrizumab, pemetrexed, carboplatin or cisplatin active ingredients and or any excipients;

18. Those who have a history of psychotropic drug abuse and can not give up or have mental disorders;

Other conditions that increase the risk associated with participating in the study or the study drug and, in the judgment of the investigator, may result in patients not suitable for inclusion in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 1 Year
  From the date Into this study to tumor progression or death for any

SECONDARY OUTCOMES:
Objective response rate | 2 Year
  it is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR.
Overall survival | 2 Year
  The time from the beginning of treatment to the death of the subject due to various reasons, calculated by the intended treatment population
Disease Control Rate | 2 Year
  the rate of CR, PR plus SD
Duration of Response | 2 Year
  Cr or PR to the first assessment of PD or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: lin Lin, doctor, Principal Investigator — Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No